CLINICAL TRIAL: NCT02320487
Title: A Phase II, Open-Label Study of Obinutuzumab Plus Bendamustine (BG) in Patients With Previously Untreated Chronic Lymphocytic Leukemia
Brief Title: A Study of Obinutuzumab + Bendamustine (BG) in Participants With Previously Untreated Chronic Lymphocytic Leukemia (CLL)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Genentech, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ML29538
Record Dates: First submitted 2014-12-16; First posted 2014-12-19 (Estimated); Results first posted 2017-12-21 (Actual); Last update posted 2020-02-11 (Actual); Status verified 2020-02

CONDITIONS: Chronic Lymphocytic Leukemia
MeSH Terms: conditions — Leukemia, Lymphocytic, Chronic, B-Cell | interventions — Bendamustine Hydrochloride; obinutuzumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Obinutuzumab + Bendamustine (BG) (Experimental): Participants received obinutuzumab + bendamustine (BG) induction therapy in 28-day cycles for 6 cycles.
  Interventions: Drug: Bendamustine; Drug: Obinutuzumab

INTERVENTIONS:
Drug: Bendamustine — Bendamustine was administered as an intravenous infusion at a dose of 90 milligrams per square meter (mg/m^2) on Days 2 and 3 Cycle 1; and on Days 1 and 2 Cycles 2-6.
  Other Names: Treanda; Levact
Drug: Obinutuzumab — Obinutuzumab was administered as an intravenous infusion at a dose of 100 milligrams (mg) on Day 1 Cycle 1; at a dose of 900 mg on Day 2 Cycle 1; at a dose of 1000 mg on Days 8 and 15 Cycle 1, and Day 1 Cycles 2-6.
  Other Names: GA101; Gazyva™; RO5072759

SUMMARY:
This is a Phase 2, open-label, multicenter study to evaluate the safety and efficacy of BG induction therapy in participants with previously untreated CLL. The anticipated time on study treatment is 24 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Participants must satisfy one of the criteria for treatment initiation, as outlined in the iwCLL NCI-WG guidelines. The criteria include: (a) Evidence of progressive marrow failure as manifested by the development of, or worsening of, anemia and/or thrombocytopenia, (b) Massive (i.e., greater than or equal to [>=] 6 centimeters [cm] below the left costal margin) or progressive or symptomatic splenomegaly, (c) Massive nodes (i.e., >= 10 cm in longest diameter) or progressive or symptomatic lymphadenopathy, (d) Progressive lymphocytosis with an increase of greater than (>) 50 percent (%) over a 2-month period or lymphocyte doubling time (LDT) of less than (<) 6 months, (e) Autoimmune anemia and/or thrombocytopenia that is poorly responsive to corticosteroids or other standard therapy, (f) Constitutional symptoms, defined as any one or more of the following disease-related symptoms or signs: unintentional weight loss of >=10% within the previous 6 months, significant fatigue (i.e., Eastern Cooperative Oncology Group Performance Status [ECOG PS] of 2 or worse or the inability to work or perform usual activities), fevers higher than 100.5 degrees Fahrenheit (°F)/38.0 degrees Celsius (°C) for >= 2 weeks without other evidence of infection, or night sweats for >1 month without evidence of infection
* Absolute neutrophil count (ANC) >=1.5 × 10^9 per liter (/L) and platelets >=75 × 10^9/L unless cytopenia is caused by the underlying disease, i.e., no evidence of additional bone marrow dysfunction (e.g., myelodysplastic syndrome, hypoplastic bone marrow)
* Life expectancy >6 months
* ECOG PS of 0, 1, or 2
* Willing to use acceptable contraceptive measures as defined by the protocol during and at least for 6 months (male participants) or 12 months (female participants) after the last dose of study drug

Exclusion Criteria:

* Pregnant or lactating, or intending to become pregnant during the study: Women who are not postmenopausal (>=12 months of non-therapy-induced amenorrhea) or surgically sterile must have a negative serum pregnancy test result within 14 days prior to initiation of study drug
* Participants who have received previous CLL therapy, including investigational therapies
* Transformation of CLL to aggressive non-Hodgkin's lymphoma (Richter's transformation)
* Inadequate renal function
* Inadequate liver function: National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) Grade 3 liver function tests (aspartate aminotransferase [AST] or alanine aminotransferase [ALT] >5× upper limit of normal [ULN] for >2 weeks; bilirubin >3× ULN) unless due to underlying disease
* History of other malignancy, which could affect compliance with the protocol or interpretation of results
* Participants with active bacterial, viral, or fungal infection requiring systemic treatment
* Participants with known infection with human immunodeficiency virus (HIV) or human T-cell leukemia virus 1 (HTLV-1)
* Positive hepatitis serology: (a) Participants with positive serology for hepatitis B, defined as positivity for hepatitis B surface antigen (HBsAg), or participants who are HBsAg negative but are hepatitis B core antibody (anti-HBc) positive, (b) Participants positive for anti-HBc, but with negative hepatitis B Virus (HBV) deoxyribonucleic acid (DNA), will be considered for inclusion by the Medical Monitor on a case-by-case basis in order to ensure feasibility of monthly DNA testing and availability of appropriate care in case of hepatitis B reactivation, (c) Participants with positive serology for hepatitis C (HCV) unless HCV (by ribonucleic acid [RNA]) is confirmed negative
* History of severe allergic or anaphylactic reactions to monoclonal antibodies
* Evidence of significant, uncontrolled concomitant diseases that could affect compliance with the protocol or interpretation of results, including significant cardiovascular disease (such as New York Heart Association Class III or IV cardiac disease, myocardial infarction within the previous 6 months, unstable arrhythmias, or unstable angina) or pulmonary disease (including obstructive pulmonary disease and history of symptomatic bronchospasm)
* Vaccination with a live vaccine a minimum of 30 days prior to study treatment
* Use of investigational agents of any kind within 30 days before study treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 102 (Actual)
Dates: Start 2015-03-31 (Actual); Primary Completion 2016-11-07 (Actual); Study Completion 2019-02-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (26):
- United States (26):
  - Clearview Cancer Institute, Huntsville, Alabama
  - Southern Cancer Center - Mobile, Mobile, Alabama
  - Ironwood Cancer TX & Rsch Ctrs, Chandler, Arizona
  - Arizona Oncology Associates, PC - HAL, Tempe, Arizona
  - Arizona Oncology Associates, PC - HOPE, Tucson, Arizona
  - Highlands Oncology Group, Fayetteville, Arkansas
  - Rocky Mountain Cancer Center - Aurora, Aurora, Colorado
  - Cancer Care and Hematology, Fort Collins, Colorado
  - Piedmont Cancer Institute, PC, Atlanta, Georgia
  - Northwest Georgia Oncology Centers PC - Marietta, Marietta, Georgia
  - Cancer Care & Hematology; Specialists of Chicagoland, Niles, Illinois
  - Fort Wayne Med Oncology & Hematology Inc, Fort Wayne, Indiana
  - Center For Cancer and Blood Disorders, Bethesda, Maryland
  - Regional Cancer Care Associates LLC - Morristown, Morristown, New Jersey
  - San Juan Oncology Associates, Farmington, New Mexico
  - Stony Brook University Hospital, Stony Brook, New York
  - Northwest Cancer Specialists - Portland (N Broadway), Portland, Oregon
  - Oregon Health and Science University, Portland, Oregon
  - Willamette Valley Cancer Insitute and Research Center, Springfield, Oregon
  - Texas Oncology-Arlington, Arlington, Texas
  - Texas Oncology-Tyler, Irving, Texas
  - Joe Arrington Cancer Research & Treatment Center, Lubbock, Texas
  - Cancer Care Centers of South Texas-HOAST - San Antonio, New Braunfels, Texas
  - Northern Utah Associates, Ogden, Utah
  - Virginia Cancer Specialists, PC, Fairfax, Virginia
  - Yakima Valley Memorial Hospital/North Star Lodge, Yakima, Washington

REFERENCES:
- [Derived] Sharman JP, Burke JM, Yimer HA, Boxer MA, Babu S, Li J, Mun Y, Danilov AV; GIBB study investigators. Phase 2, multicenter GIBB study of obinutuzumab plus bendamustine in previously untreated patients with chronic lymphocytic leukemia. Leuk Lymphoma. 2021 Apr;62(4):791-800. doi: 10.1080/10428194.2020.1850719. Epub 2020 Nov 26. PMID 33243049

RESULTS

PARTICIPANT FLOW:
Groups:
- Obinutuzumab + Bendamustine (BG): Participants received obinutuzumab + bendamustine (BG) therapy in 28-day cycles for 6 cycles.
Period: Overall Study
Arm/Group | Obinutuzumab + Bendamustine (BG)
Started | 102
Completed | 81 (Completed = completed the 6-cycle Treatment Period.)
Not Completed | 21
Not completed — Reason not Specified | 1
Not completed — Physician Decision | 5
Not completed — Withdrawal by Subject | 1
Not completed — Death | 3
Not completed — Adverse Event | 11

BASELINE CHARACTERISTICS:
Arm/Group | Obinutuzumab + Bendamustine (BG)
Number analyzed (Participants) | 102
Age, Continuous [Mean (Standard Deviation); unit: years] | 62.5 (10.79)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 32
  Male | 70
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 97
  Unknown or Not Reported | 4
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 2
  White | 98
  More than one race | 0
  Unknown or Not Reported | 2

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Complete Response (CR), as Determined by the Investigator Using International Workshop on Chronic Lymphocytic Leukemia National Cancer Institute-Working Group (iwCLL NCI-WG) Guidelines
Description: The CR rate was defined as CR or CR with incomplete blood count recovery (CRi), assessed by the investigator according to iwCLL NCI-WG criteria. The definition of confirmed CR required all of the following criteria as assessed at least 2 months after completion of therapy: peripheral blood lymphocytes < 4 times 10^9 cells/L; absence of significant lymphadenopathy, hepatomegaly, or splenomegaly due to CLL involvement; absence of constitutional symptoms; normal complete blood count (CBC) without need for transfusion or exogenous growth factors, as exhibited by neutrophils >/= 1.5 times 10^9 cells/L, platelets > 100 times 10^9 cells/L, and hemoglobin > 11.0 g/dL; normocellular BM aspirate with < 30% lymphocytes; absence of lymphoid nodules; and BM biopsy without CLL activity. Those fulfilling CR criteria but who have persistent anemia, thrombocytopenia, or neutropenia were considered CRi.
Time Frame: 2 to 3 months after the last infusion of study treatment (up to approximately 228 to 258 days)
Population: The modified intent-to-treat (mITT) population included enrolled participants who received at least one dose of BG.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Obinutuzumab + Bendamustine (BG)
Number analyzed (Participants) | 102
percentage of participants | 50.0 [39.9 to 60.1]

2. Secondary Outcome: Percentage of Participants With Objective Response of CR or Partial Response (PR) at the End of Induction Therapy, as Determined by the Investigator Using iwCLL NCI-WG Guidelines
Description: CR is defined in the previous outcome measure. The definition of PR required that the following be documented for minimum 2 months: >/= 50% decrease in peripheral blood lymphocytes from Baseline; reduction in lymphadenopathy; >/= 50% reduction in spleen or liver enlargement; and CBC with one of the following without need for transfusion or exogenous growth factors: polymorphonuclear leukocytes >/= 1.5 times 10^9 cells/L, platelets > 100 times 10^9 cells/L or >/= 50% improvement from Baseline, or hemoglobin > 11.0 g/dL or >/= 50% improvement from Baseline.
Time Frame: 2 to 3 months after the last infusion of study treatment (up to approximately 228 to 258 days)
Population: The mITT population included enrolled participants who received at least one dose of BG.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Obinutuzumab + Bendamustine (BG)
Number analyzed (Participants) | 102
percentage of participants | 89.2 [81.5 to 94.5]

3. Secondary Outcome: Duration of Response Among Participants With Objective Response of CR or PR, as Determined by the Investigator Using iwCLL NCI-WG Guidelines
Description: Duration of response was defined as the time from the first assessment of CR, CRi, PR, or nodular partial response (nPR) to the first documentation of PD or death, whichever occurred first. CR, CRi, and PR are identified in previous outcome measures. Participants with lymphoid nodules who otherwise met CR criteria were considered nPR. Participants with post-baseline response assessments (excluding progressive disease) but with no end-of-induction treatment response available were censored on Day 1, and those with end-of-induction treatment response available but who did not experience death or disease progression before the end of the study were censored on the day of the last available assessment.
Time Frame: From the first assessment of CR, CRi, PR, or nPR (at up to approximately 228 to 258 days) until disease progression, relapse, or death from any cause, whichever occurred first (up to 46 months)
Population: The mITT population included enrolled participants who received at least one dose of BG. Analysis performed for participants with response.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Obinutuzumab + Bendamustine (BG)
Number analyzed (Participants) | 91
months | NA [NA to NA] — Not estimable due to the low number participants with events that qualified for the analysis.

4. Secondary Outcome: Progression-Free Survival (PFS), as Determined by the Investigator Using iwCLL NCI-WG Guidelines
Description: PFS was defined as the time from the start of induction treatment (Day 1) to the first occurrence of disease progression, relapse as determined by the investigator using iwCLL NCI WG guidelines, or death (within 28 days after the last dose of study drug), whichever occurred first. Disease progression: at least one of the following: lymphadenopathy; increase in the liver or spleen size by 50% or more or the appearance of hepatomegaly or splenomegaly; an increase in the number of blood lymphocytes by 50% or more with at least 5000 B lymphocytes per microliter; transformation to a more aggressive histology; occurrence of cytopenia (neutropenia, anemia, or thrombocytopenia) attributable to CLL. Relapse: Having achieved CR or PR, but after a period of 6 or more months, having demonstrated evidence of disease progression. Participants who did not experience death or disease progression before the end of the study were censored on the day of the last available assessment.
Time Frame: Day 1 until disease progression, relapse, or death from any cause, whichever occurred first (up to 46 months)
Population: The mITT population included enrolled participants who received at least one dose of BG.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Obinutuzumab + Bendamustine (BG)
Number analyzed (Participants) | 102
months | NA [35.0 to NA] — Not estimable due to the low number participants with events that qualified for the analysis.

5. Secondary Outcome: Overall Survival (OS)
Description: OS was defined as the time from the start of induction treatment to death from any cause. Participants who did not experience death or disease progression before the end of the study were censored on the day of the last available assessment.
Time Frame: Day 1 until death from any cause (up to 46 months)
Population: The mITT population included enrolled participants who received at least one dose of BG.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Obinutuzumab + Bendamustine (BG)
Number analyzed (Participants) | 102
months | NA [NA to NA] — Not estimable due to the low number participants with events that qualified for the analysis.

6. Secondary Outcome: Percentage of Participants Who Achieved Minimal Residual Disease (MRD)-Negative Status in Bone Marrow at Any Time During the Study
Description: MRD was assessed by 4-color flow cytometry, using iwCLL criteria for MRD negativity (<1 CLL cell detected in 10,000 leukocytes) in bone marrow aspirate. Flow cytometry provides rapid analysis of multiple characteristics of single cells by using light to count and profile cells in a fluid mixture.
Time Frame: Up to 46 months
Population: The mITT population included enrolled participants who received at least one dose of BG. Data are reported for evaluable participants.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Obinutuzumab + Bendamustine (BG)
Number analyzed (Participants) | 51
percentage of participants | 58.8 [44.2 to 72.4]

7. Secondary Outcome: Percentage of Participants Who Achieved MRD-Negative Status in Peripheral Blood at Any Time During the Study
Description: MRD was assessed by 4-color flow cytometry, using iwCLL criteria for MRD negativity (<1 CLL cell detected in 10,000 leukocytes) in peripheral blood. Flow cytometry provides rapid analysis of multiple characteristics of single cells by using light to count and profile cells in a fluid mixture.
Time Frame: Baseline up to 46 months
Population: as for outcome 6
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Obinutuzumab + Bendamustine (BG)
Number analyzed (Participants) | 95
percentage of participants | 83.2 [74.1 to 90.1]

8. Secondary Outcome: Time to MRD-Negative Status in Peripheral Blood
Description: MRD was assessed by 4-color flow cytometry, using iwCLL criteria for MRD negativity if the value is <10^-4 (<1 CLL cell detected in 10,000 leukocytes) in peripheral blood. Flow cytometry provides rapid analysis of multiple characteristics of single cells by using light to count and profile cells in a fluid mixture. Time to MRD-negative status is defined as the time between MRD positivity (>= 10^-4) or the time of first dose treatment for patients who were missing MRD status assessment at baseline to the first achievement of MRD negativity in the peripheral blood.
Time Frame: Baseline up to 46 months
Population: The mITT population included enrolled participants who received at least one dose of BG.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Obinutuzumab + Bendamustine (BG)
Number analyzed (Participants) | 102
months | 8.2 [7.1 to 10.3]

9. Secondary Outcome: Duration of MRD-Negativity in Peripheral Blood Among Participants Who Achieved MRD-Negative Status
Description: MRD was assessed by 4-color flow cytometry, using iwCLL criteria for MRD negativity (<1 CLL cell detected in 10,000 leukocytes) in peripheral blood. Flow cytometry provides rapid analysis of multiple characteristics of single cells by using light to count and profile cells in a fluid mixture. Duration of MRD-negativity among patients who achieved MRD negativity in the study is defined as the period between the first occurrence of MRD-negative status and a subsequent MRD-positive status.
Time Frame: Baseline up to 46 months
Population: as for outcome 6
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Obinutuzumab + Bendamustine (BG)
Number analyzed (Participants) | 79
months | 28.9 [23.0 to NA] — Not estimable due to the low number of participants with events that qualified for the analysis.

10. Secondary Outcome: Minimum Observed Concentration (Ctrough) of Obinutuzumab After Cycle 2
Description: Ctrough is the measured concentration of a drug at the end of a dosing interval at steady state.
Time Frame: Pre-infusion (0 hours) on Day 1 Cycle 3 (1 cycle = 28 days)
Population: The PK (pharmacokinetic) Evaluable Population included all ITT participants in the study who received any dose of study drug (obinutuzumab or bendamustine) and had at least one PK assessment. Data are reported for evaluable participants.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanograms per milliliter (ng/mL)
Arm/Group | Obinutuzumab + Bendamustine (BG)
Number analyzed (Participants) | 95
nanograms per milliliter (ng/mL) | 235.92 (48.01)

11. Secondary Outcome: Ctrough of Obinutuzumab After Cycle 4
Description: Ctrough is the measured concentration of a drug at the end of a dosing interval at steady state.
Time Frame: Pre-infusion (0 hours) on Day 1 Cycle 5 (1 cycle = 28 days)
Population: as for outcome 10
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanograms per milliliter (ng/mL)
Arm/Group | Obinutuzumab + Bendamustine (BG)
Number analyzed (Participants) | 80
nanograms per milliliter (ng/mL) | 264.27 (46.45)

12. Secondary Outcome: Change From Baseline in the European Organisation for Research and Treatment of Cancer (EORTC) Quality of Life Questionnaire-Core 30 (QLQ-C30) Score
Description: The EORTC QLQ-C30 included global health status, functional scales (physical, role, emotional, cognitive, and social), symptom scales (fatigue, nausea/vomiting, and pain) and single items (dyspnoea, insomnia, appetite loss, constipation, diarrhea, and financial difficulties). Most questions used a 4-point scale (1 'Not at all' to 4 'Very much'; 2 questions used 7-point scale [1 'very poor' to 7 'Excellent']). Scores were averaged and transformed to 0 - 100 scale, whereby higher scores indicate greater functioning, greater quality of life, or a greater degree of symptoms, with changes of 5 - 10 points considered to be a minimally important difference to participants. A positive change from Day 1, Cycle 1 (baseline) indicates improvement. EOT=end of treatment.
Time Frame: Day 1 Cycles 1 (baseline), 3, 6; end of treatment, 2 months after last dose, every 3 months thereafter for 2 years (up to 46 months) (1 cycle = 28 days)
Population: The PRO (patient-reported outcome) Evaluable Population included all ITT participants in the study who received any dose of study treatment (obinutuzumab or bendamustine) and had both a non-missing baseline and at least one post-baseline PRO assessment. Data were not collected for the second year of follow up.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Obinutuzumab + Bendamustine (BG)
Number analyzed (Participants) | 98
score on a scale
  Global Health Status (GHS)/QoL: Cycle 3: number analyzed (Participants) | 85
  Global Health Status (GHS)/QoL: Cycle 3 | 4.02 (21.540)
  GHS/QoL: Cycle 6: number analyzed (Participants) | 76
  GHS/QoL: Cycle 6 | 5.26 (22.478)
  GHS/QoL: EOT/Early Discontinuation: number analyzed (Participants) | 79
  GHS/QoL: EOT/Early Discontinuation | 5.17 (26.731)
  GHS/QoL: Response Visit: number analyzed (Participants) | 85
  GHS/QoL: Response Visit | 10.98 (21.715)
  GHS/QoL: 3-Month Follow-Up: number analyzed (Participants) | 74
  GHS/QoL: 3-Month Follow-Up | 10.25 (24.733)
  GHS/QoL: 6-Month Follow-Up: number analyzed (Participants) | 66
  GHS/QoL: 6-Month Follow-Up | 5.68 (30.140)
  GHS/QoL: 9-Month Follow-Up: number analyzed (Participants) | 72
  GHS/QoL: 9-Month Follow-Up | 9.26 (23.384)
  GHS/QoL: 12-Month Follow-Up: number analyzed (Participants) | 79
  GHS/QoL: 12-Month Follow-Up | 6.43 (24.676)
  GHS/QoL: 15-Month Follow-Up: number analyzed (Participants) | 71
  GHS/QoL: 15-Month Follow-Up | 6.57 (25.969)
  GHS/QoL: 18-Month Follow-Up: number analyzed (Participants) | 72
  GHS/QoL: 18-Month Follow-Up | 9.84 (26.732)
  GHS/QoL: 21-Month Follow-Up: number analyzed (Participants) | 68
  GHS/QoL: 21-Month Follow-Up | 7.60 (27.117)
  GHS/QoL: 24-Month Follow-Up: number analyzed (Participants) | 58
  GHS/QoL: 24-Month Follow-Up | 8.91 (27.388)
  GHS/QoL: 27-Month Follow-Up: number analyzed (Participants) | 49
  GHS/QoL: 27-Month Follow-Up | 13.26 (24.468)
  GHS/QoL: 30-Month Follow-Up: number analyzed (Participants) | 5
  GHS/QoL: 30-Month Follow-Up | 1.66 (28.501)
  Physical Function: Cycle 3: number analyzed (Participants) | 86
  Physical Function: Cycle 3 | -2.46 (14.948)
  Physical Function: Cycle 6: number analyzed (Participants) | 77
  Physical Function: Cycle 6 | 0.00 (12.842)
  Phys. Function: EOT/Early Discontinuation: number analyzed (Participants) | 79
  Phys. Function: EOT/Early Discontinuation | 2.62 (15.188)
  Physical Function: Response Visit: number analyzed (Participants) | 85
  Physical Function: Response Visit | 3.90 (14.705)
  Physical Function: 3-Month Follow-Up: number analyzed (Participants) | 74
  Physical Function: 3-Month Follow-Up | 4.14 (13.769)
  Physical Function: 6-Month Follow-Up: number analyzed (Participants) | 66
  Physical Function: 6-Month Follow-Up | 1.62 (17.308)
  Physical Function: 9-Month Follow-Up: number analyzed (Participants) | 72
  Physical Function: 9-Month Follow-Up | 4.95 (15.208)
  Physical Function: 12-Month Follow-Up: number analyzed (Participants) | 80
  Physical Function: 12-Month Follow-Up | 3.00 (15.221)
  Physical Function: 15-Month Follow-Up: number analyzed (Participants) | 71
  Physical Function: 15-Month Follow-Up | 2.44 (17.647)
  Physical Function: 18-Month Follow-Up: number analyzed (Participants) | 72
  Physical Function: 18-Month Follow-Up | 1.11 (18.589)
  Physical Function: 21-Month Follow-Up: number analyzed (Participants) | 68
  Physical Function: 21-Month Follow-Up | 1.37 (13.509)
  Physical Function: 24-Month Follow-Up: number analyzed (Participants) | 58
  Physical Function: 24-Month Follow-Up | 3.10 (14.467)
  Physical Function: 27-Month Follow-Up: number analyzed (Participants) | 49
  Physical Function: 27-Month Follow-Up | 4.22 (14.057)
  Physical Function: 30-Month Follow-Up: number analyzed (Participants) | 5
  Physical Function: 30-Month Follow-Up | 5.34 (8.691)
  Role Function: Cycle 3: number analyzed (Participants) | 86
  Role Function: Cycle 3 | 6.01 (24.775)
  Role Function: Cycle 6: number analyzed (Participants) | 77
  Role Function: Cycle 6 | 4.11 (27.193)
  Role Function: EOT/Early Discontinuation: number analyzed (Participants) | 79
  Role Function: EOT/Early Discontinuation | 10.55 (27.108)
  Role Function: Response Visit: number analyzed (Participants) | 85
  Role Function: Response Visit | 13.14 (29.106)
  Role Function: 3-Month Follow-Up: number analyzed (Participants) | 74
  Role Function: 3-Month Follow-Up | 14.87 (28.210)
  Role Function: 6-Month Follow-Up: number analyzed (Participants) | 66
  Role Function: 6-Month Follow-Up | 10.86 (29.453)
  Role Function: 9-Month Follow-Up: number analyzed (Participants) | 72
  Role Function: 9-Month Follow-Up | 15.51 (27.312)
  Role Function: 12-Month Follow-Up: number analyzed (Participants) | 80
  Role Function: 12-Month Follow-Up | 10.63 (28.591)
  Role Function: 15-Month Follow-Up: number analyzed (Participants) | 71
  Role Function: 15-Month Follow-Up | 12.68 (30.920)
  Role Function: 18-Month Follow-Up: number analyzed (Participants) | 72
  Role Function: 18-Month Follow-Up | 10.88 (33.352)
  Role Function: 21-Month Follow-Up: number analyzed (Participants) | 67
  Role Function: 21-Month Follow-Up | 10.95 (28.656)
  Role Function: 24-Month Follow-Up: number analyzed (Participants) | 58
  Role Function: 24-Month Follow-Up | 11.49 (30.780)
  Role Function: 27-Month Follow-Up: number analyzed (Participants) | 49
  Role Function: 27-Month Follow-Up | 14.97 (30.285)
  Role Function: 30-Month Follow-Up: number analyzed (Participants) | 5
  Role Function: 30-Month Follow-Up | -13.33 (36.132)
  Emotional Function: Cycle 3: number analyzed (Participants) | 85
  Emotional Function: Cycle 3 | 7.91 (18.092)
  Emotional Function: Cycle 6: number analyzed (Participants) | 76
  Emotional Function: Cycle 6 | 6.29 (18.304)
  Emotional Function: EOT/Early Discont.: number analyzed (Participants) | 79
  Emotional Function: EOT/Early Discont. | 9.60 (18.302)
  Emotional Function: Response Visit: number analyzed (Participants) | 85
  Emotional Function: Response Visit | 9.12 (18.663)
  Emotional Function: 3-Month Follow-Up: number analyzed (Participants) | 74
  Emotional Function: 3-Month Follow-Up | 8.11 (18.861)
  Emotional Function: 6-Month Follow-Up: number analyzed (Participants) | 66
  Emotional Function: 6-Month Follow-Up | 6.94 (19.424)
  Emotional Function: 9-Month Follow-Up: number analyzed (Participants) | 72
  Emotional Function: 9-Month Follow-Up | 11.00 (13.402)
  Emotional Function: 12-Month Follow-Up: number analyzed (Participants) | 79
  Emotional Function: 12-Month Follow-Up | 7.81 (18.793)
  Emotional Function: 15-Month Follow-Up: number analyzed (Participants) | 71
  Emotional Function: 15-Month Follow-Up | 6.34 (23.883)
  Emotional Function: 18-Month Follow-Up: number analyzed (Participants) | 72
  Emotional Function: 18-Month Follow-Up | 5.75 (22.214)
  Emotional Function: 21-Month Follow-Up: number analyzed (Participants) | 68
  Emotional Function: 21-Month Follow-Up | 7.11 (19.597)
  Emotional Function: 24-Month Follow-Up: number analyzed (Participants) | 58
  Emotional Function: 24-Month Follow-Up | 9.77 (19.380)
  Emotional Function: 27-Month Follow-Up: number analyzed (Participants) | 49
  Emotional Function: 27-Month Follow-Up | 10.15 (18.845)
  Emotional Function: 30-Month Follow-Up: number analyzed (Participants) | 5
  Emotional Function: 30-Month Follow-Up | 8.33 (15.591)
  Cognitive Function: Cycle 3: number analyzed (Participants) | 85
  Cognitive Function: Cycle 3 | 2.55 (22.640)
  Cognitive Function: Cycle 6: number analyzed (Participants) | 76
  Cognitive Function: Cycle 6 | -1.75 (25.177)
  Cognitive Function: EOT/Early Discont.: number analyzed (Participants) | 79
  Cognitive Function: EOT/Early Discont. | 0.42 (17.697)
  Cognitive Function: Response Visit: number analyzed (Participants) | 85
  Cognitive Function: Response Visit | 2.74 (20.387)
  Cognitive Function: 3-Month Follow-Up: number analyzed (Participants) | 74
  Cognitive Function: 3-Month Follow-Up | 2.25 (17.946)
  Cognitive Function: 6-Month Follow-Up: number analyzed (Participants) | 66
  Cognitive Function: 6-Month Follow-Up | 1.77 (23.043)
  Cognitive Function: 9-Month Follow-Up: number analyzed (Participants) | 72
  Cognitive Function: 9-Month Follow-Up | 6.02 (17.312)
  Cognitive Function: 12-Month Follow-Up: number analyzed (Participants) | 79
  Cognitive Function: 12-Month Follow-Up | 1.48 (19.646)
  Cognitive Function: 15-Month Follow-Up: number analyzed (Participants) | 71
  Cognitive Function: 15-Month Follow-Up | 2.11 (20.878)
  Cognitive Function: 18-Month Follow-Up: number analyzed (Participants) | 72
  Cognitive Function: 18-Month Follow-Up | 2.55 (20.105)
  Cognitive Function: 21-Month Follow-Up: number analyzed (Participants) | 68
  Cognitive Function: 21-Month Follow-Up | 3.19 (20.815)
  Cognitive Function: 24-Month Follow-Up: number analyzed (Participants) | 58
  Cognitive Function: 24-Month Follow-Up | 4.02 (18.550)
  Cognitive Function: 27-Month Follow-Up: number analyzed (Participants) | 49
  Cognitive Function: 27-Month Follow-Up | 1.70 (16.401)
  Cognitive Function: 30-Month Follow-Up: number analyzed (Participants) | 5
  Cognitive Function: 30-Month Follow-Up | -3.33 (21.726)
  Social Function: Cycle 3: number analyzed (Participants) | 85
  Social Function: Cycle 3 | -2.35 (21.386)
  Social Function: Cycle 6: number analyzed (Participants) | 76
  Social Function: Cycle 6 | -4.17 (23.590)
  Social Function: EOT/Early Discontinuation: number analyzed (Participants) | 79
  Social Function: EOT/Early Discontinuation | 2.53 (23.279)
  Social Function: Response Visit: number analyzed (Participants) | 85
  Social Function: Response Visit | 5.69 (24.874)
  Social Function: 3-Month Follow-Up: number analyzed (Participants) | 74
  Social Function: 3-Month Follow-Up | 5.41 (23.587)
  Social Function: 6-Month Follow-Up: number analyzed (Participants) | 66
  Social Function: 6-Month Follow-Up | -0.25 (26.872)
  Social Function: 9-Month Follow-Up: number analyzed (Participants) | 72
  Social Function: 9-Month Follow-Up | 8.10 (19.579)
  Social Function: 12-Month Follow-Up: number analyzed (Participants) | 79
  Social Function: 12-Month Follow-Up | 2.74 (24.667)
  Social Function: 15-Month Follow-Up: number analyzed (Participants) | 71
  Social Function: 15-Month Follow-Up | 3.76 (25.696)
  Social Function: 18-Month Follow-Up: number analyzed (Participants) | 72
  Social Function: 18-Month Follow-Up | 3.70 (27.296)
  Social Function: 21-Month Follow-Up: number analyzed (Participants) | 68
  Social Function: 21-Month Follow-Up | 2.70 (26.952)
  Social Function: 24-Month Follow-Up: number analyzed (Participants) | 58
  Social Function: 24-Month Follow-Up | 5.46 (21.032)
  Social Function: 27-Month Follow-Up: number analyzed (Participants) | 49
  Social Function: 27-Month Follow-Up | 7.48 (23.088)
  Social Function: 30-Month Follow-Up: number analyzed (Participants) | 5
  Social Function: 30-Month Follow-Up | -10.00 (30.277)
  Fatigue: Cycle 3: number analyzed (Participants) | 86
  Fatigue: Cycle 3 | -4.01 (25.433)
  Fatigue: Cycle 6: number analyzed (Participants) | 77
  Fatigue: Cycle 6 | -5.48 (24.558)
  Fatigue: EOT/Early Discontinuation: number analyzed (Participants) | 79
  Fatigue: EOT/Early Discontinuation | -11.67 (24.324)
  Fatigue: Response Visit: number analyzed (Participants) | 85
  Fatigue: Response Visit | -16.34 (25.291)
  Fatigue: 3-Month Follow-Up: number analyzed (Participants) | 74
  Fatigue: 3-Month Follow-Up | -15.92 (24.266)
  Fatigue: 6-Month Follow-Up: number analyzed (Participants) | 66
  Fatigue: 6-Month Follow-Up | -13.64 (24.171)
  Fatigue: 9-Month Follow-Up: number analyzed (Participants) | 72
  Fatigue: 9-Month Follow-Up | -17.28 (23.947)
  Fatigue: 12-Month Follow-Up: number analyzed (Participants) | 80
  Fatigue: 12-Month Follow-Up | -13.12 (24.261)
  Fatigue: 15-Month Follow-Up: number analyzed (Participants) | 71
  Fatigue: 15-Month Follow-Up | -11.27 (25.441)
  Fatigue: 18-Month Follow-Up: number analyzed (Participants) | 72
  Fatigue: 18-Month Follow-Up | -13.43 (24.946)
  Fatigue: 21-Month Follow-Up: number analyzed (Participants) | 68
  Fatigue: 21-Month Follow-Up | -13.07 (22.465)
  Fatigue: 24-Month Follow-Up: number analyzed (Participants) | 58
  Fatigue: 24-Month Follow-Up | -14.37 (21.429)
  Fatigue: 27-Month Follow-Up: number analyzed (Participants) | 49
  Fatigue: 27-Month Follow-Up | -14.51 (23.373)
  Fatigue: 30-Month Follow-Up: number analyzed (Participants) | 5
  Fatigue: 30-Month Follow-Up | -2.22 (16.480)
  Nausea/Vomiting: Cycle 3: number analyzed (Participants) | 86
  Nausea/Vomiting: Cycle 3 | 2.33 (16.990)
  Nausea/Vomiting: Cycle 6: number analyzed (Participants) | 77
  Nausea/Vomiting: Cycle 6 | 3.68 (14.210)
  Nausea/Vomiting: EOT/Early Discontinuation: number analyzed (Participants) | 79
  Nausea/Vomiting: EOT/Early Discontinuation | 2.32 (13.273)
  Nausea/Vomiting: Response Visit: number analyzed (Participants) | 85
  Nausea/Vomiting: Response Visit | -0.39 (15.209)
  Nausea/Vomiting: 3-Month Follow-Up: number analyzed (Participants) | 74
  Nausea/Vomiting: 3-Month Follow-Up | -1.58 (9.624)
  Nausea/Vomiting: 6-Month Follow-Up: number analyzed (Participants) | 66
  Nausea/Vomiting: 6-Month Follow-Up | -1.26 (12.164)
  Nausea/Vomiting: 9-Month Follow-Up: number analyzed (Participants) | 72
  Nausea/Vomiting: 9-Month Follow-Up | -0.23 (16.428)
  Nausea/Vomiting: 12-Month Follow-Up: number analyzed (Participants) | 80
  Nausea/Vomiting: 12-Month Follow-Up | -1.04 (13.350)
  Nausea/Vomiting: 15-Month Follow-Up: number analyzed (Participants) | 71
  Nausea/Vomiting: 15-Month Follow-Up | 0.70 (13.926)
  Nausea/Vomiting: 18-Month Follow-Up: number analyzed (Participants) | 72
  Nausea/Vomiting: 18-Month Follow-Up | -0.23 (13.267)
  Nausea/Vomiting: 21-Month Follow-Up: number analyzed (Participants) | 68
  Nausea/Vomiting: 21-Month Follow-Up | -1.72 (13.240)
  Nausea/Vomiting: 24-Month Follow-Up: number analyzed (Participants) | 58
  Nausea/Vomiting: 24-Month Follow-Up | -2.01 (14.333)
  Nausea/Vomiting: 27-Month Follow-Up: number analyzed (Participants) | 49
  Nausea/Vomiting: 27-Month Follow-Up | -1.70 (14.925)
  Nausea/Vomiting: 30-Month Follow-Up: number analyzed (Participants) | 5
  Nausea/Vomiting: 30-Month Follow-Up | 10.00 (14.910)
  Pain: Cycle 3: number analyzed (Participants) | 86
  Pain: Cycle 3 | -3.68 (17.969)
  Pain: Cycle 6: number analyzed (Participants) | 77
  Pain: Cycle 6 | 0.65 (26.826)
  Pain: EOT/Early Discontinuation: number analyzed (Participants) | 79
  Pain: EOT/Early Discontinuation | -1.90 (21.012)
  Pain: Response Visit: number analyzed (Participants) | 85
  Pain: Response Visit | -4.90 (20.865)
  Pain: 3-Month Follow-Up: number analyzed (Participants) | 74
  Pain: 3-Month Follow-Up | -1.80 (17.570)
  Pain: 6-Month Follow-Up: number analyzed (Participants) | 66
  Pain: 6-Month Follow-Up | -1.52 (20.615)
  Pain: 9-Month Follow-Up: number analyzed (Participants) | 72
  Pain: 9-Month Follow-Up | -0.69 (20.448)
  Pain: 12-Month Follow-Up: number analyzed (Participants) | 80
  Pain: 12-Month Follow-Up | -0.21 (24.947)
  Pain: 15-Month Follow-Up: number analyzed (Participants) | 71
  Pain: 15-Month Follow-Up | 0.94 (26.709)
  Pain: 18-Month Follow-Up: number analyzed (Participants) | 72
  Pain: 18-Month Follow-Up | -0.46 (25.326)
  Pain: 21-Month Follow-Up: number analyzed (Participants) | 68
  Pain: 21-Month Follow-Up | -0.00 (23.035)
  Pain: 24-Month Follow-Up: number analyzed (Participants) | 58
  Pain: 24-Month Follow-Up | -2.59 (19.447)
  Pain: 27-Month Follow-Up: number analyzed (Participants) | 49
  Pain: 27-Month Follow-Up | -5.44 (26.654)
  Pain: 30-Month Follow-Up: number analyzed (Participants) | 5
  Pain: 30-Month Follow-Up | 6.67 (48.015)
  Dyspnoea: Cycle 3: number analyzed (Participants) | 86
  Dyspnoea: Cycle 3 | 0.39 (27.294)
  Dyspnoea: Cycle 6: number analyzed (Participants) | 77
  Dyspnoea: Cycle 6 | -1.73 (25.874)
  Dyspnoea: EOT/Early Discontinuation: number analyzed (Participants) | 79
  Dyspnoea: EOT/Early Discontinuation | -5.91 (31.013)
  Dyspnoea: Response Visit: number analyzed (Participants) | 85
  Dyspnoea: Response Visit | -5.88 (30.069)
  Dyspnoea: 3-Month Follow-Up: number analyzed (Participants) | 74
  Dyspnoea: 3-Month Follow-Up | -9.46 (27.872)
  Dyspnoea: 6-Month Follow-Up: number analyzed (Participants) | 66
  Dyspnoea: 6-Month Follow-Up | -8.08 (27.463)
  Dyspnoea: 9-Month Follow-Up: number analyzed (Participants) | 72
  Dyspnoea: 9-Month Follow-Up | -7.87 (29.334)
  Dyspnoea: 12-Month Follow-Up: number analyzed (Participants) | 80
  Dyspnoea: 12-Month Follow-Up | -5.83 (30.824)
  Dyspnoea: 15-Month Follow-Up: number analyzed (Participants) | 71
  Dyspnoea: 15-Month Follow-Up | -5.63 (29.270)
  Dyspnoea: 18-Month Follow-Up: number analyzed (Participants) | 72
  Dyspnoea: 18-Month Follow-Up | -7.87 (28.796)
  Dyspnoea: 21-Month Follow-Up: number analyzed (Participants) | 68
  Dyspnoea: 21-Month Follow-Up | -8.82 (27.289)
  Dyspnoea: 24-Month Follow-Up: number analyzed (Participants) | 58
  Dyspnoea: 24-Month Follow-Up | -7.47 (28.642)
  Dyspnoea: 27-Month Follow-Up: number analyzed (Participants) | 49
  Dyspnoea: 27-Month Follow-Up | -11.56 (31.587)
  Dyspnoea: 30-Month Follow-Up: number analyzed (Participants) | 5
  Dyspnoea: 30-Month Follow-Up | -20.00 (18.256)
  Insomnia: Cycle 3: number analyzed (Participants) | 86
  Insomnia: Cycle 3 | -6.59 (27.450)
  Insomnia: Cycle 6: number analyzed (Participants) | 77
  Insomnia: Cycle 6 | -9.09 (24.565)
  Insomnia: EOT/Early Discontinuation: number analyzed (Participants) | 79
  Insomnia: EOT/Early Discontinuation | -9.70 (25.684)
  Insomnia: Response Visit: number analyzed (Participants) | 85
  Insomnia: Response Visit | -10.98 (28.354)
  Insomnia: 3-Month Follow-Up: number analyzed (Participants) | 74
  Insomnia: 3-Month Follow-Up | -9.46 (25.596)
  Insomnia: 6-Month Follow-Up: number analyzed (Participants) | 66
  Insomnia: 6-Month Follow-Up | -14.65 (29.312)
  Insomnia: 9-Month Follow-Up: number analyzed (Participants) | 72
  Insomnia: 9-Month Follow-Up | -12.50 (29.306)
  Insomnia: 12-Month Follow-Up: number analyzed (Participants) | 79
  Insomnia: 12-Month Follow-Up | -9.70 (31.193)
  Insomnia: 15-Month Follow-Up: number analyzed (Participants) | 71
  Insomnia: 15-Month Follow-Up | -13.61 (30.643)
  Insomnia: 18-Month Follow-Up: number analyzed (Participants) | 72
  Insomnia: 18-Month Follow-Up | -8.80 (30.640)
  Insomnia: 21-Month Follow-Up: number analyzed (Participants) | 68
  Insomnia: 21-Month Follow-Up | -7.84 (29.991)
  Insomnia: 24-Month Follow-Up: number analyzed (Participants) | 58
  Insomnia: 24-Month Follow-Up | -14.37 (28.691)
  Insomnia: 27-Month Follow-Up: number analyzed (Participants) | 49
  Insomnia: 27-Month Follow-Up | -10.20 (36.136)
  Insomnia: 30-Month Follow-Up: number analyzed (Participants) | 5
  Insomnia: 30-Month Follow-Up | -6.67 (49.443)
  Appetite Loss: Cycle 3: number analyzed (Participants) | 86
  Appetite Loss: Cycle 3 | -2.71 (20.589)
  Appetite Loss: Cycle 6: number analyzed (Participants) | 77
  Appetite Loss: Cycle 6 | 0.00 (26.490)
  Appetite Loss: EOT/Early Discontinuation: number analyzed (Participants) | 79
  Appetite Loss: EOT/Early Discontinuation | -3.80 (18.480)
  Appetite Loss: Response Visit: number analyzed (Participants) | 85
  Appetite Loss: Response Visit | -7.06 (21.878)
  Appetite Loss: 3-Month Follow-Up: number analyzed (Participants) | 74
  Appetite Loss: 3-Month Follow-Up | -9.91 (18.896)
  Appetite Loss: 6-Month Follow-Up: number analyzed (Participants) | 66
  Appetite Loss: 6-Month Follow-Up | -9.60 (18.270)
  Appetite Loss: 9-Month Follow-Up: number analyzed (Participants) | 71
  Appetite Loss: 9-Month Follow-Up | -10.80 (22.378)
  Appetite Loss: 12-Month Follow-Up: number analyzed (Participants) | 80
  Appetite Loss: 12-Month Follow-Up | -8.75 (20.364)
  Appetite Loss: 15-Month Follow-Up: number analyzed (Participants) | 71
  Appetite Loss: 15-Month Follow-Up | -6.57 (24.312)
  Appetite Loss: 18-Month Follow-Up: number analyzed (Participants) | 72
  Appetite Loss: 18-Month Follow-Up | -7.41 (19.557)
  Appetite Loss: 21-Month Follow-Up: number analyzed (Participants) | 68
  Appetite Loss: 21-Month Follow-Up | -4.90 (23.928)
  Appetite Loss: 24-Month Follow-Up: number analyzed (Participants) | 58
  Appetite Loss: 24-Month Follow-Up | -7.47 (20.748)
  Appetite Loss: 27-Month Follow-Up: number analyzed (Participants) | 49
  Appetite Loss: 27-Month Follow-Up | -8.16 (19.872)
  Appetite Loss: 30-Month Follow-Up: number analyzed (Participants) | 5
  Appetite Loss: 30-Month Follow-Up | -6.67 (14.906)
  Constipation: Cycle 3: number analyzed (Participants) | 85
  Constipation: Cycle 3 | 3.92 (34.661)
  Constipation: Cycle 6: number analyzed (Participants) | 76
  Constipation: Cycle 6 | -0.00 (24.944)
  Constipation: EOT/Early Discontinuation: number analyzed (Participants) | 78
  Constipation: EOT/Early Discontinuation | -4.27 (18.105)
  Constipation: Response Visit: number analyzed (Participants) | 84
  Constipation: Response Visit | -4.36 (24.147)
  Constipation: 3-Month Follow-Up: number analyzed (Participants) | 73
  Constipation: 3-Month Follow-Up | -5.02 (18.979)
  Constipation: 6-Month Follow-Up: number analyzed (Participants) | 66
  Constipation: 6-Month Follow-Up | -6.06 (19.312)
  Constipation: 9-Month Follow-Up: number analyzed (Participants) | 71
  Constipation: 9-Month Follow-Up | -5.16 (24.975)
  Constipation: 12-Month Follow-Up: number analyzed (Participants) | 79
  Constipation: 12-Month Follow-Up | -3.80 (25.028)
  Constipation: 15-Month Follow-Up: number analyzed (Participants) | 71
  Constipation: 15-Month Follow-Up | -3.76 (19.147)
  Constipation: 18-Month Follow-Up: number analyzed (Participants) | 72
  Constipation: 18-Month Follow-Up | -0.46 (24.059)
  Constipation: 21-Month Follow-Up: number analyzed (Participants) | 68
  Constipation: 21-Month Follow-Up | -2.45 (22.538)
  Constipation: 24-Month Follow-Up: number analyzed (Participants) | 58
  Constipation: 24-Month Follow-Up | -6.32 (21.134)
  Constipation: 27-Month Follow-Up: number analyzed (Participants) | 49
  Constipation: 27-Month Follow-Up | -6.80 (21.494)
  Constipation: 30-Month Follow-Up: number analyzed (Participants) | 5
  Constipation: 30-Month Follow-Up | 0.00 (0.000)
  Diarrhoea: Cycle 3: number analyzed (Participants) | 85
  Diarrhoea: Cycle 3 | 1.18 (21.483)
  Diarrhoea: Cycle 6: number analyzed (Participants) | 76
  Diarrhoea: Cycle 6 | 4.82 (24.767)
  Diarrhoea: EOT/Early Discontinuation: number analyzed (Participants) | 79
  Diarrhoea: EOT/Early Discontinuation | 4.64 (29.105)
  Diarrhoea: Response Visit: number analyzed (Participants) | 85
  Diarrhoea: Response Visit | 2.75 (24.780)
  Diarrhoea: 3-Month Follow-Up: number analyzed (Participants) | 74
  Diarrhoea: 3-Month Follow-Up | -2.25 (20.886)
  Diarrhoea: 6-Month Follow-Up: number analyzed (Participants) | 66
  Diarrhoea: 6-Month Follow-Up | -1.01 (24.085)
  Diarrhoea: 9-Month Follow-Up: number analyzed (Participants) | 72
  Diarrhoea: 9-Month Follow-Up | 3.24 (23.174)
  Diarrhoea: 12-Month Follow-Up: number analyzed (Participants) | 78
  Diarrhoea: 12-Month Follow-Up | -0.43 (21.816)
  Diarrhoea: 15-Month Follow-Up: number analyzed (Participants) | 71
  Diarrhoea: 15-Month Follow-Up | 0.00 (25.197)
  Diarrhoea: 18-Month Follow-Up: number analyzed (Participants) | 72
  Diarrhoea: 18-Month Follow-Up | -2.78 (26.090)
  Diarrhoea: 21-Month Follow-Up: number analyzed (Participants) | 68
  Diarrhoea: 21-Month Follow-Up | 3.43 (28.875)
  Diarrhoea: 24-Month Follow-Up: number analyzed (Participants) | 58
  Diarrhoea: 24-Month Follow-Up | -0.57 (22.067)
  Diarrhoea: 27-Month Follow-Up: number analyzed (Participants) | 49
  Diarrhoea: 27-Month Follow-Up | 1.36 (21.471)
  Diarrhoea: 30-Month Follow-Up: number analyzed (Participants) | 5
  Diarrhoea: 30-Month Follow-Up | 0.00 (23.568)
  Financial Difficulty: Cycle 3: number analyzed (Participants) | 85
  Financial Difficulty: Cycle 3 | 0.78 (25.186)
  Financial Difficulty: Cycle 6: number analyzed (Participants) | 76
  Financial Difficulty: Cycle 6 | -2.19 (27.934)
  Financial Difficulty: EOT/Early Discont.: number analyzed (Participants) | 79
  Financial Difficulty: EOT/Early Discont. | -1.27 (26.923)
  Financial Difficulty: Response Visit: number analyzed (Participants) | 85
  Financial Difficulty: Response Visit | -3.53 (29.107)
  Financial Difficulty: 3-Month Follow-Up: number analyzed (Participants) | 74
  Financial Difficulty: 3-Month Follow-Up | -5.86 (27.784)
  Financial Difficulty: 6-Month Follow-Up: number analyzed (Participants) | 65
  Financial Difficulty: 6-Month Follow-Up | -7.18 (27.947)
  Financial Difficulty: 9-Month Follow-Up: number analyzed (Participants) | 71
  Financial Difficulty: 9-Month Follow-Up | -7.04 (26.972)
  Financial Difficulty: 12-Month Follow-Up: number analyzed (Participants) | 79
  Financial Difficulty: 12-Month Follow-Up | -3.80 (30.188)
  Financial Difficulty: 15-Month Follow-Up: number analyzed (Participants) | 71
  Financial Difficulty: 15-Month Follow-Up | -8.45 (29.125)
  Financial Difficulty: 18-Month Follow-Up: number analyzed (Participants) | 72
  Financial Difficulty: 18-Month Follow-Up | -6.02 (31.313)
  Financial Difficulty: 21-Month Follow-Up: number analyzed (Participants) | 68
  Financial Difficulty: 21-Month Follow-Up | -6.86 (25.471)
  Financial Difficulty: 24-Month Follow-Up: number analyzed (Participants) | 58
  Financial Difficulty: 24-Month Follow-Up | -7.47 (26.523)
  Financial Difficulty: 27-Month Follow-Up: number analyzed (Participants) | 49
  Financial Difficulty: 27-Month Follow-Up | -11.56 (31.587)
  Financial Difficulty: 30-Month Follow-Up: number analyzed (Participants) | 5
  Financial Difficulty: 30-Month Follow-Up | -13.33 (29.813)

13. Secondary Outcome: Change From Baseline in the EORTC Quality of Life Questionnaire-Chronic Lymphocytic Leukemia 16 (QLQ-CLL16) Score
Description: The EORTC Quality of Life Questionnaire-Chronic Lymphocytic Leukemia 16 (QLQ-CLL16) module included assessments of fatigue, treatment side effects, disease symptoms, infection, social activities, and future health worries. Final scores are transformed such that they range from 0 - 100, whereby higher scores indicate greater functioning, greater quality of life, or a greater degree of symptoms, with changes of 5 - 10 points considered to be a minimally important difference to participants. A positive change from Day 1, Cycle 1 (baseline) indicates improvement. EOT=end of treatment.
Time Frame: as for outcome 12
Population: The PRO Evaluable Population included all ITT participants in the study who received any dose of study treatment (obinutuzumab or bendamustine) and had both a non-missing baseline and at least one post-baseline PRO assessment. Data were not collected for the second year of follow up.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Obinutuzumab + Bendamustine (BG)
Number analyzed (Participants) | 98
score on a scale
  Fatigue: Cycle 3: number analyzed (Participants) | 86
  Fatigue: Cycle 3 | -12.02 (26.892)
  Fatigue: Cycle 6: number analyzed (Participants) | 77
  Fatigue: Cycle 6 | -10.17 (26.373)
  Fatigue: EOT/Early Discontinuation: number analyzed (Participants) | 79
  Fatigue: EOT/Early Discontinuation | -12.87 (30.306)
  Fatigue: Response Visit: number analyzed (Participants) | 84
  Fatigue: Response Visit | -21.23 (30.759)
  Fatigue: 3-Month Follow-Up: number analyzed (Participants) | 74
  Fatigue: 3-Month Follow-Up | -20.04 (29.323)
  Fatigue: 6-Month Follow-Up: number analyzed (Participants) | 65
  Fatigue: 6-Month Follow-Up | -17.44 (25.418)
  Fatigue: 9-Month Follow-Up: number analyzed (Participants) | 71
  Fatigue: 9-Month Follow-Up | -22.77 (27.780)
  Fatigue: 12-Month Follow-Up: number analyzed (Participants) | 77
  Fatigue: 12-Month Follow-Up | -17.32 (25.569)
  Fatigue: 15-Month Follow-Up: number analyzed (Participants) | 70
  Fatigue: 15-Month Follow-Up | -14.52 (30.153)
  Fatigue: 18-Month Follow-Up: number analyzed (Participants) | 71
  Fatigue: 18-Month Follow-Up | -15.49 (30.122)
  Fatigue: 21-Month Follow-Up: number analyzed (Participants) | 67
  Fatigue: 21-Month Follow-Up | -16.42 (28.646)
  Fatigue: 24-Month Follow-Up: number analyzed (Participants) | 56
  Fatigue: 24-Month Follow-Up | -24.70 (25.621)
  Fatigue: 27-Month Follow-Up: number analyzed (Participants) | 46
  Fatigue: 27-Month Follow-Up | -19.56 (26.597)
  Fatigue: 30-Month Follow-Up: number analyzed (Participants) | 5
  Fatigue: 30-Month Follow-Up | -6.67 (53.489)
  Side Effects: Cycle 3: number analyzed (Participants) | 86
  Side Effects: Cycle 3 | 1.52 (12.019)
  Side Effects: Cycle 6: number analyzed (Participants) | 77
  Side Effects: Cycle 6 | 0.07 (16.072)
  Side Effects: EOT/Early Discontinuation: number analyzed (Participants) | 79
  Side Effects: EOT/Early Discontinuation | -0.67 (16.357)
  Side Effects: Response Visit: number analyzed (Participants) | 84
  Side Effects: Response Visit | -2.08 (14.520)
  Side Effects: 3-Month Follow-Up: number analyzed (Participants) | 74
  Side Effects: 3-Month Follow-Up | -3.30 (12.904)
  Side Effects: 6-Month Follow-Up: number analyzed (Participants) | 65
  Side Effects: 6-Month Follow-Up | -2.61 (15.182)
  Side Effects: 9-Month Follow-Up: number analyzed (Participants) | 71
  Side Effects: 9-Month Follow-Up | -3.36 (14.548)
  Side Effects: 12-Month Follow-Up: number analyzed (Participants) | 77
  Side Effects: 12-Month Follow-Up | -2.27 (14.841)
  Side Effects: 15-Month Follow-Up: number analyzed (Participants) | 70
  Side Effects: 15-Month Follow-Up | -3.17 (14.355)
  Side Effects: 18-Month Follow-Up: number analyzed (Participants) | 71
  Side Effects: 18-Month Follow-Up | -4.54 (14.813)
  Side Effects: 21-Month Follow-Up: number analyzed (Participants) | 67
  Side Effects: 21-Month Follow-Up | -1.66 (16.277)
  Side Effects: 24-Month Follow-Up: number analyzed (Participants) | 56
  Side Effects: 24-Month Follow-Up | -3.08 (13.699)
  Side Effects: 27-Month Follow-Up: number analyzed (Participants) | 46
  Side Effects: 27-Month Follow-Up | -2.96 (14.434)
  Side Effects: 30-Month Follow-Up: number analyzed (Participants) | 5
  Side Effects: 30-Month Follow-Up | -11.67 (4.566)
  Disease Symptoms: Cycle 3: number analyzed (Participants) | 86
  Disease Symptoms: Cycle 3 | -9.56 (18.196)
  Disease Symptoms: Cycle 6: number analyzed (Participants) | 77
  Disease Symptoms: Cycle 6 | -8.30 (20.039)
  Disease Symptoms: EOT/Early Discontinuation: number analyzed (Participants) | 79
  Disease Symptoms: EOT/Early Discontinuation | -10.02 (20.371)
  Disease Symptoms: Response Visit: number analyzed (Participants) | 84
  Disease Symptoms: Response Visit | -12.67 (18.019)
  Disease Symptoms: 3-Month Follow-Up: number analyzed (Participants) | 74
  Disease Symptoms: 3-Month Follow-Up | -12.20 (18.630)
  Disease Symptoms: 6-Month Follow-Up: number analyzed (Participants) | 65
  Disease Symptoms: 6-Month Follow-Up | -10.13 (16.699)
  Disease Symptoms: 9-Month Follow-Up: number analyzed (Participants) | 71
  Disease Symptoms: 9-Month Follow-Up | -12.28 (18.478)
  Disease Symptoms: 12-Month Follow-Up: number analyzed (Participants) | 77
  Disease Symptoms: 12-Month Follow-Up | -8.62 (18.297)
  Disease Symptoms: 15-Month Follow-Up: number analyzed (Participants) | 70
  Disease Symptoms: 15-Month Follow-Up | -9.05 (19.284)
  Disease Symptoms: 18-Month Follow-Up: number analyzed (Participants) | 71
  Disease Symptoms: 18-Month Follow-Up | -10.41 (20.632)
  Disease Symptoms: 21-Month Follow-Up: number analyzed (Participants) | 67
  Disease Symptoms: 21-Month Follow-Up | -9.16 (21.398)
  Disease Symptoms: 24-Month Follow-Up: number analyzed (Participants) | 56
  Disease Symptoms: 24-Month Follow-Up | -10.71 (17.675)
  Disease Symptoms: 27-Month Follow-Up: number analyzed (Participants) | 46
  Disease Symptoms: 27-Month Follow-Up | -11.41 (19.904)
  Disease Symptoms: 30-Month Follow-Up: number analyzed (Participants) | 5
  Disease Symptoms: 30-Month Follow-Up | -5.00 (20.917)
  Infection: Cycle 3: number analyzed (Participants) | 86
  Infection: Cycle 3 | 6.20 (18.182)
  Infection: Cycle 6: number analyzed (Participants) | 77
  Infection: Cycle 6 | 4.11 (16.406)
  Infection: EOT/Early Discontinuation: number analyzed (Participants) | 79
  Infection: EOT/Early Discontinuation | 1.65 (15.199)
  Infection: Response Visit: number analyzed (Participants) | 84
  Infection: Response Visit | 0.76 (17.528)
  Infection: 3-Month Follow-Up: number analyzed (Participants) | 74
  Infection: 3-Month Follow-Up | 2.59 (20.779)
  Infection: 6-Month Follow-Up: number analyzed (Participants) | 65
  Infection: 6-Month Follow-Up | 3.46 (23.611)
  Infection: 9-Month Follow-Up: number analyzed (Participants) | 71
  Infection: 9-Month Follow-Up | 1.45 (17.135)
  Infection: 12-Month Follow-Up: number analyzed (Participants) | 78
  Infection: 12-Month Follow-Up | 4.42 (22.269)
  Infection: 15-Month Follow-Up: number analyzed (Participants) | 70
  Infection: 15-Month Follow-Up | 2.86 (19.602)
  Infection: 18-Month Follow-Up: number analyzed (Participants) | 71
  Infection: 18-Month Follow-Up | 2.62 (22.532)
  Infection: 21-Month Follow-Up: number analyzed (Participants) | 67
  Infection: 21-Month Follow-Up | 2.78 (18.502)
  Infection: 24-Month Follow-Up: number analyzed (Participants) | 56
  Infection: 24-Month Follow-Up | 0.89 (15.134)
  Infection: 27-Month Follow-Up: number analyzed (Participants) | 46
  Infection: 27-Month Follow-Up | 1.45 (14.731)
  Infection: 30-Month Follow-Up: number analyzed (Participants) | 5
  Infection: 30-Month Follow-Up | -5.00 (9.502)
  Social Activities: Cycle 3: number analyzed (Participants) | 85
  Social Activities: Cycle 3 | -3.92 (28.827)
  Social Activities: Cycle 6: number analyzed (Participants) | 76
  Social Activities: Cycle 6 | -3.95 (34.412)
  Social Activities: EOT/Early Discont.: number analyzed (Participants) | 78
  Social Activities: EOT/Early Discont. | -6.41 (33.141)
  Social Activities: Response Visit: number analyzed (Participants) | 83
  Social Activities: Response Visit | -9.24 (33.054)
  Social Activities: 3-Month Follow-Up: number analyzed (Participants) | 73
  Social Activities: 3-Month Follow-Up | -11.87 (27.983)
  Social Activities: 6-Month Follow-Up: number analyzed (Participants) | 64
  Social Activities: 6-Month Follow-Up | -4.69 (33.527)
  Social Activities: 9-Month Follow-Up: number analyzed (Participants) | 70
  Social Activities: 9-Month Follow-Up | -13.33 (28.033)
  Social Activities: 12-Month Follow-Up: number analyzed (Participants) | 76
  Social Activities: 12-Month Follow-Up | -7.89 (27.145)
  Social Activities: 15-Month Follow-Up: number analyzed (Participants) | 69
  Social Activities: 15-Month Follow-Up | -6.76 (34.099)
  Social Activities: 18-Month Follow-Up: number analyzed (Participants) | 70
  Social Activities: 18-Month Follow-Up | -5.71 (31.583)
  Social Activities: 21-Month Follow-Up: number analyzed (Participants) | 66
  Social Activities: 21-Month Follow-Up | -4.55 (32.495)
  Social Activities: 24-Month Follow-Up: number analyzed (Participants) | 55
  Social Activities: 24-Month Follow-Up | -11.51 (28.845)
  Social Activities: 27-Month Follow-Up: number analyzed (Participants) | 46
  Social Activities: 27-Month Follow-Up | -9.42 (29.534)
  Social Activities: 30-Month Follow-Up: number analyzed (Participants) | 5
  Social Activities: 30-Month Follow-Up | 0.00 (66.668)
  Future Health Worries: Cycle 3: number analyzed (Participants) | 83
  Future Health Worries: Cycle 3 | -20.08 (30.329)
  Future Health Worries: Cycle 6: number analyzed (Participants) | 76
  Future Health Worries: Cycle 6 | -14.04 (29.946)
  Future Health Worries: EOT/Early Discont.: number analyzed (Participants) | 79
  Future Health Worries: EOT/Early Discont. | -18.57 (32.794)
  Future Health Worries: Response Visit: number analyzed (Participants) | 84
  Future Health Worries: Response Visit | -20.24 (28.351)
  Future Health Worries: 3-Month Follow-Up: number analyzed (Participants) | 73
  Future Health Worries: 3-Month Follow-Up | -25.11 (29.805)
  Future Health Worries: 6-Month Follow-Up: number analyzed (Participants) | 65
  Future Health Worries: 6-Month Follow-Up | -17.44 (30.680)
  Future Health Worries: 9-Month Follow-Up: number analyzed (Participants) | 71
  Future Health Worries: 9-Month Follow-Up | -23.47 (27.253)
  Future Health Worries: 12-Month Follow-Up: number analyzed (Participants) | 78
  Future Health Worries: 12-Month Follow-Up | -19.23 (26.053)
  Future Health Worries: 15-Month Follow-Up: number analyzed (Participants) | 70
  Future Health Worries: 15-Month Follow-Up | -17.14 (33.929)
  Future Health Worries: 18-Month Follow-Up: number analyzed (Participants) | 71
  Future Health Worries: 18-Month Follow-Up | -19.72 (34.540)
  Future Health Worries: 21-Month Follow-Up: number analyzed (Participants) | 66
  Future Health Worries: 21-Month Follow-Up | -21.21 (27.820)
  Future Health Worries: 24-Month Follow-Up: number analyzed (Participants) | 55
  Future Health Worries: 24-Month Follow-Up | -21.82 (30.911)
  Future Health Worries: 27-Month Follow-Up: number analyzed (Participants) | 46
  Future Health Worries: 27-Month Follow-Up | -25.36 (31.572)
  Future Health Worries: 30-Month Follow-Up: number analyzed (Participants) | 5
  Future Health Worries: 30-Month Follow-Up | -6.67 (27.892)

14. Secondary Outcome: Number of Hospitalizations Due to Adverse Events (AEs)
Description: An AE is any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease temporally associated with the use of a study drug, whether or not considered related to the study drug.
Time Frame: Day 1 up to 46 months
Population: The safety population included participants who received any amount of study treatment.
Measure: Mean (Standard Deviation); unit: hospitalizations
Arm/Group | Obinutuzumab + Bendamustine (BG)
Number analyzed (Participants) | 102
hospitalizations | 1.43 (0.634)

15. Secondary Outcome: Percentage of Participants With Adverse Events (AEs)
Description: as for outcome 14
Time Frame: Day 1 up to 46 months
Population: The safety population included participants who received any amount of study treatment.
Measure: Number; unit: percentage of participants
Arm/Group | Obinutuzumab + Bendamustine (BG)
Number analyzed (Participants) | 102
percentage of participants | 100

ADVERSE EVENTS:
Time Frame: Day 1 up to 46 months
Arm/Group | Obinutuzumab + Bendamustine (BG)
All-Cause Mortality (participants affected / at risk) | 7/102
Serious Adverse Events (participants affected / at risk) | 31/102
Other Adverse Events (participants affected / at risk) | 101/102
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Obinutuzumab + Bendamustine (BG) (N=102)
Febrile neutropenia (Blood and lymphatic system disorders) | 4 (4)
Anaemia (Blood and lymphatic system disorders) | 1 (1)
Cardiac arrest (Cardiac disorders) | 1 (1)
Myocardial infarction (Cardiac disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (1)
Pyrexia (General disorders) | 5 (5)
Pneumonia (Infections and infestations) | 7 (8)
Urinary tract infection (Infections and infestations) | 2 (2)
Catheter site infection (Infections and infestations) | 1 (1)
Infection (Infections and infestations) | 1 (1)
Oesophageal candidiasis (Infections and infestations) | 1 (1)
Septic shock (Infections and infestations) | 1 (1)
Infusion related reaction (Injury, poisoning and procedural complications) | 2 (2)
Blood creatinine increased (Investigations) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 3 (3)
Tumour lysis syndrome (Metabolism and nutrition disorders) | 4 (4)
Failure to thrive (Metabolism and nutrition disorders) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Hypotension (Vascular disorders) | 2 (2)
Cardiac failure congestive (Cardiac disorders) | 1 (1)
Progressive multifocal leukoencephalopathy (Infections and infestations) | 1 (1)
Sepsis (Infections and infestations) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Obinutuzumab + Bendamustine (BG) (N=102)
Neutropenia (Blood and lymphatic system disorders) | 36 (53)
Thrombocytopenia (Blood and lymphatic system disorders) | 20 (42)
Anaemia (Blood and lymphatic system disorders) | 14 (18)
Nausea (Gastrointestinal disorders) | 54 (74)
Constipation (Gastrointestinal disorders) | 27 (29)
Diarrhoea (Gastrointestinal disorders) | 24 (34)
Vomiting (Gastrointestinal disorders) | 21 (33)
Abdominal pain (Gastrointestinal disorders) | 11 (13)
Dyspepsia (Gastrointestinal disorders) | 7 (7)
Fatigue (General disorders) | 36 (48)
Pyrexia (General disorders) | 35 (44)
Oedema peripheral (General disorders) | 16 (16)
Chills (General disorders) | 13 (13)
Upper respiratory tract infection (Infections and infestations) | 14 (15)
Bronchitis (Infections and infestations) | 6 (6)
Infusion related reaction (Injury, poisoning and procedural complications) | 76 (96)
Neutrophil count decreased (Investigations) | 15 (24)
Platelet count decreased (Investigations) | 8 (15)
Weight decreased (Investigations) | 8 (10)
Dehydration (Metabolism and nutrition disorders) | 15 (18)
Decreased appetite (Metabolism and nutrition disorders) | 12 (13)
Hypokalaemia (Metabolism and nutrition disorders) | 9 (14)
Hypomagnesaemia (Metabolism and nutrition disorders) | 6 (7)
Hyponatraemia (Metabolism and nutrition disorders) | 6 (6)
Arthralgia (Musculoskeletal and connective tissue disorders) | 13 (16)
Bone pain (Musculoskeletal and connective tissue disorders) | 8 (8)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 9 (10)
Back pain (Musculoskeletal and connective tissue disorders) | 7 (7)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 7 (7)
Headache (Nervous system disorders) | 19 (24)
Dizziness (Nervous system disorders) | 12 (16)
Dysgeusia (Nervous system disorders) | 8 (8)
Insomnia (Psychiatric disorders) | 19 (20)
Anxiety (Psychiatric disorders) | 7 (7)
Cough (Respiratory, thoracic and mediastinal disorders) | 17 (21)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 8 (8)
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 6 (8)
Rash (Skin and subcutaneous tissue disorders) | 28 (42)
Dry skin (Skin and subcutaneous tissue disorders) | 10 (10)
Pruritus (Skin and subcutaneous tissue disorders) | 7 (10)
Night sweats (Skin and subcutaneous tissue disorders) | 6 (6)
Flushing (Vascular disorders) | 7 (9)
Hypotension (Vascular disorders) | 8 (8)
Pneumonia (Infections and infestations) | 6 (6)
Myalgia (Musculoskeletal and connective tissue disorders) | 7 (8)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.